CLINICAL TRIAL: NCT06702215
Title: Cortical Plasticity of the Tactile Mirror System in Borderline Personality Disorder
Acronym: SG2019-EXP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Agnese Zazio, Researcher, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SG2019-EXP2; SG-2019-12370473 (Other Grant/Funding Number: Italian Ministry of Health (Ricerca 'Finalizzata 2019'))
Record Dates: First submitted 2024-11-15; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: transcranial magnetic stimulation; brain plasticity; paired associative stimulation; somatosensory domain; mirror neuron system; borderline personality disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Clinical Protocols; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Both patients with BPD and healthy controls will undergo two experimental conditions, in counterbalanced order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental cm-PAS protocol followed by control cm-PAS protocol (Experimental): Participants will undergo the experimental cm-PAS protocol in the first session of the experiment, followed by the control cm-PAS protocol in the second session. The experimental and the control PAS protocols will differ in the timing of TMS delivery, one effective and the other one uneffective in inducing plastic effects, as shown by previous studies on healthy participants.
  Interventions: Device: Cross-modal paired associative stimulation (cm-PAS) protocol
- Control cm-PAS protocol followed by experimental cm-PAS protocol (Experimental): Participants will undergo the control cm-PAS protocol in the first session of the experiment, followed by the experimental cm-PAS protocol in the second session. The experimental and the control PAS protocols will differ in the timing of TMS delivery, one effective and the other one uneffective in inducing plastic effects, as shown by previous studies on healthy participants.
  Interventions: Device: Cross-modal paired associative stimulation (cm-PAS) protocol

INTERVENTIONS:
Device: Cross-modal paired associative stimulation (cm-PAS) protocol — The cross-modal Paired Associative Stimulation (cm-PAS) will consist of a visual stimulus depicting a hand being touched repeatedly paired with a transcranial magnetic stimulation (TMS) pulse delivered over the right primary somatosensory area, for a total of 150 paired stimuli delivered at a fixed frequency of 0.1 Hz. The time interval between the visual-touch onset and the TMS pulse will be 20 ms for the experimental session and 100 ms for the control session.
  Other Names: PAS; TMS; transcranial magnetic stimulation

SUMMARY:
People with borderline personality disorder (BPD) show alterations in the empathic abilities, which may involve the functioning of the mirror neuron system in the somatosensory domain. In the so-called Tactile Mirror System, the observation of a touch on someone else's body activates a cortical network also involved in tactile perception, including the primary somatosensory cortex. While alterations of mirror-like systems have been suggested in BPD, plasticity mechanisms within these systems are underexplored.

The present study aims to shed light on the possible neurophysiological alterations within the Tactile Mirror System in people with BPD, employing a non-invasive transcranial magnetic stimulation protocol, called cross-modal paired associative stimulation (cm-PAS), to induce brain plasticity.

DETAILED DESCRIPTION:
While previous studies have suggested mirror system alterations in BPD, still little is known about the integrity of a basic neurophysiological mechanism such as brain plasticity within these systems. Considering that the development of mentalization and empathic abilities appears to rely on early associative learning and metaplasticity, it has been suggested that the pathophysiology of BPD may be associated with alterations in neuronal plasticity, mediated by N-methyl-D-aspartate (NMDA) neurotransmission; however, evidence is still lacking. Importantly, the integrity of plasticity mechanisms may represent a critical factor for the effectiveness of therapeutic interventions.

Paired associative stimulation (PAS) protocols represent a well-established tool to non-invasively induce brain plasticity effects in humans. To induce changes in synaptic efficacy, PAS protocols exploit the Hebbian learning rule and the concept of spike-timing dependent plasticity observed at the cellular level, namely that neural connections are strengthened (or weakened) in the case of repeated activations of the presynaptic neuron before the postsynaptic neuron (or vice-versa) in a critical time interval of a few tens of ms. In classical PAS protocols targeting the somatosensory system (S1-PAS), a peripheral electrical stimulus over the wrist (acting as presynaptic activation) is repeatedly paired with a transcranial magnetic stimulation (TMS) pulse over S1 in the contralateral hemisphere (acting as postsynaptic activation). Depending on the time interval between the two stimuli, the S1-PAS may induce long-term potentiation or depression (LTP- or LTD-like, respectively) effects, lasting up to 30 minutes after protocol delivery. In addition to neurophysiological effects (i.e., somatosensory evoked potential modulation), these plastic mechanisms have also been detected by exploiting behavioral measures of S1 functioning, such as tactile acuity.

PAS protocols have also been used to target multisensory integration networks: here, the peripheral and cortical stimuli belong to different systems. Recently, a cross-modal PAS (cm-PAS) has been developed in the visuo-tactile domain, with the aim of targeting the Tactile Mirror System. Compared to classical S1-PAS, in cm-PAS the peripheral electrical stimulus on the wrist is replaced by a visual stimulus of a hand being touched. The efficacy of the cm-PAS in inducing LTP-like mechanisms has been shown in a series of experiments, consisting of an increase in tactile acuity that was specific for the time interval between the visual stimulus and the TMS, for the site of cortical stimulation, and for the content of the visual stimulus. Moreover, cm-PAS modulated a neurophysiological correlate of S1 activity, namely, the amplitude of the P40 component of somatosensory-evoked potentials increased after cm-PAS. Overall, these findings are consistent with the hypothesis that when seeing a human touch on someone else's body, S1 is recruited by mirror-like mechanisms and can be involved in plasticity mechanisms.

Taking together the existing evidence, the present study aims to shed light on the neural basis of interpersonal dysfunction in BPD by bridging the gap between the literature on empathic alterations in BPD patients on the one hand and on the neurophysiological underpinnings of TaMS and its plastic properties in the healthy population on the other hand. Specifically, the integrity of plastic modulations within the Tactile Mirror System will be investigated in BPD patients, by employing the previously described cm-PAS.

The present study will involve BPD 24 patients and 24 healthy controls (HCs) undergoing two sessions of cm-PAS, i.e., an experimental session and a control session. BPD patients will be matched one-to-one with HCs for gender and age. The two groups will be compared in the cognitive dimensions of empathic abilities, measured by means of a self-report questionnaire (Questionnaire for Cognitive and Affective Empathy). To assess the effects of the cm-PAS, both groups will undergo a behavioral task involving visuo-tactile stimuli, before and after the cm-PAS protocol, and performance will be evaluated in terms of accuracy and reaction times.

ELIGIBILITY:
Inclusion Criteria:

* All participants: right handedness (Edinburgh Handedness Inventory; Oldfield, 1971)
* Patients group: clinical diagnosis of BPD. The severity of the symptoms will be assessed by means of the Zanarini rating scale for BPD (ZAN-BPD, Zanarini, 2003) and the Symptoms Check-list 90 Revised (SCL-90-R, Derogatis, 1994). Depressive symptoms will be evaluated with the Beck Depression Inventory II (BDI-II, Beck, 1988), impulsiveness with the Barratt Impulsiveness Scale (BIS, Patton, Stanford, & Barratt, 1995), and alexithymia with the Toronto Alexithymia Scale (TAS-20, Bagby, Taylor, & Parker, 1994). Moreover, interpersonal functioning will be evaluated with the Interpersonal Problems (IIP, Pilkonis, Kim, Proietti, & Barkham, 1996), and attachment style will be assessed with the Attachment Style Questionnaire (Feeney, Noller, & Hanrahan, 1994). Finally, the Childhood Trauma Questionnaire (CTQ; Bernstein & Fink, 1998) will be administered for the assessment of traumatic experiences, and the Inventory of statements about self-injury (ISAS, Klonsky & Glenn, 2009) for the evaluation of self-harm.

Exclusion Criteria:

* All participants: Contraindication to TMS (Rossi et al., 2021)
* All participants: Anamnesis or evidence of any central nervous system alteration
* Patients group: Comorbidity with schizophrenia and other psychotic disorders, according to DSM-5, and in case of unstable pharmacological therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Visuo-tactile performance | Within 30 minutes before and after the cm-PAS protocol in each experimental session
  Behavioral performance will be obtained from an adapted version of the visuo-tactile spatial congruency task, already used in previous studies to investigate the tactile mirror system. In this task, pictures of a left and a right hand are presented on a screen in egocentric perspective, then, another hand in allocentric perspective appears on the screen and touches either the left or the right hand (i.e., visual touch). At the same time, participants receive a real touch on the left or the right hand, which can be spatially congruent or incongruent with respect to the visual touch. Participants will be asked to report the location of the real touch, i.e., on the left or on the right hand, as fast and accurately as possible, by pressing one of two buttons on a computer keyboard. Both reaction reaction times and accuracy will be considered as outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
* Behavioral performance (accuracy, reaction times) at the visuo-tactile spatial congruity task, before and after the experimental and the control cm-PAS protocol;
  * Empathic levels as indexed by self-report questionnaire
Supporting Information: Analytic Code
Time Frame: Upon acceptance of the scientific paper on study outcome.

REFERENCES:
- [Background] Zazio A, Guidali G, Maddaluno O, Miniussi C, Bolognini N. Hebbian associative plasticity in the visuo-tactile domain: A cross-modal paired associative stimulation protocol. Neuroimage. 2019 Nov 1;201:116025. doi: 10.1016/j.neuroimage.2019.116025. Epub 2019 Jul 17. PMID 31325642